CLINICAL TRIAL: NCT07133100
Title: Intrasubject Evaluation of Upper Limb Movement Precision Using the AuReha System in Individuals With Unilateral Motor Impairment
Brief Title: Evaluating Upper Limb Movement Precision With AuReha in People With One-Sided Motor Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DigitalRehab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DigitalRehab_01_2025
Record Dates: First submitted 2025-08-08; First posted 2025-08-20 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Shoulder Posterior Instability; Shoulder Anterior Instability; Shoulder Anterior Latarjet Instability; Adhesive Capsulitis, Shoulder; Prostheses
Keywords: wearable medical device; upper limb rehabilitation; inertial measurement sensors; monitoring system; supporting system; shoulder rehabilitation
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: The study has a two-arm intra-patient design, as the comparison will be made within the same subject between the healthy limb and the affected limb.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients affected by orthopedic shoulder conditions such as posterior instability, ant (Experimental): The clinical investigation is designed as an interventional, controlled, two-arm intra-patient, non-randomized study aimed at evaluating the capabilities of the AuReha system in detecting the accuracy of upper limb movements in patients with unilateral proprioceptive deficits. The comparison will be conducted within the same subject between the healthy limb and the affected limb, through the performance of proprioceptive exercises in open kinetic chain. No therapeutic or diagnostic interventions will be administered, as this is a non-invasive study focused on system validation and user feedback.
  Interventions: Device: Upper limb rehabilitation wearable device

INTERVENTIONS:
Device: Upper limb rehabilitation wearable device — The intervention consists in using the AuReha system to perform a series of upper limb rehabilitation exercises. No therapeutic or diagnostic interventions will be administered, as this is a non-invasive study focused on system validation and user feedback.

SUMMARY:
The clinical investigation is designed as a controlled, two-arm, intra-patient, non-randomized interventional study aimed at assessing the capabilities of the AuReha system in detecting upper limb movement precision in patients with unilateral proprioceptive impairment. The comparison will be conducted within the same subject, between the healthy limb and the impaired limb, through the execution of proprioceptive exercises in an open kinetic chain. The biomechanical parameters collected will include movement precision, trunk stability, compensatory movements, and joint range of motion. In addition to the quantitative analysis, qualitative data will also be collected regarding usability, wearability, and user experience of the system through questionnaires administered to both patients and healthcare professionals.

The study will be conducted at the Shoulder Team Outpatient Clinic in Forlì, enrolling approximately 52 patients.

DETAILED DESCRIPTION:
The primary goal of this clinical investigation is to support the CE certification process of the AuReha system, a wearable medical device designed for monitoring upper limb movement during rehabilitation.

Specifically, the study aims to assess the movement precision of the upper limb in individuals with unilateral motor impairment. The main objective is to compare, within the same individual, the movement accuracy of the healthy arm versus the impaired arm during a series of rehabilitation exercises guided by the AuReha system.

Secondary objectives include:

* Evaluating the usability of the AuReha system in clinical practice from the perspective of healthcare professionals using the Healthcare Systems Usability Scale (HSUS) and additional targeted questions.
* Assessing patients' user experience during proprioceptive exercises, through the System Usability Scale (SUS), the User Engagement Scale - Short Form (UES-SF), and other custom questions.
* Characterizing the wearability of the device by matching shirt sizes with patients' anthropometric measurements, using both direct observations and questionnaires.
* Analyzing the movement data collected during a specific reaching task prompted by the AuReha system, to gain deeper insight into the quality and precision of the movement performed.

These aspects aim to demonstrate the system's ability to support an optimized rehabilitation process. AuReha is designed to help patients perform their prescribed rehabilitation exercises correctly while collecting detailed biomechanical data. This allows clinicians to closely monitor the patient's response to therapy and make data-driven decisions throughout the recovery process.

ELIGIBILITY:
Inclusion Criteria:

* patients with a healthy contralateral limb
* patients affected by orthopedic shoulder conditions such as posterior instability, anterior instability, anterior Latarjet instability, adhesive capsulitis, or prostheses
* age ≥18 years
* patients who consent to participate in the study by signing the informed consent form

Exclusion Criteria:

* Pregnant and/or breastfeeding women (verified through self-declaration)
* Epilepsy
* Allergy or hypersensitivity to materials used in the medical device, specifically: polypropylene and lycra (fabric), nylon (integrated zipper), viscose and elastane (zipper integration fabric)
* Chronic headache under treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the intra-subject difference in movement accuracy during a target-reaching exercise proposed by the AuReha system, between the healthy limb and the limb affected by motor deficit | Day 1
  Unit of measurement: Percentage (%) - Movement accuracy, expressed as a percentage, measures how precisely the patient performs the prescribed movements, by assessing the deviation of the executed movement from the ideal movement to be performed.

SECONDARY OUTCOMES:
Characterization of AuReha in measuring trunk stability | Day 1
  Trunk stability is a parameter calculated by the AuReha Web Platform that assesses the inclination of the trunk across the three reference planes (frontal, sagittal, and transverse) during exercise execution. Trunk stability is an essential parameter to ensure the correct performance of upper limb movements and to prevent harmful compensations that could negatively impact recovery.
  Unit of Measure: Percentage (%)
Characterization of AuReha in measuring limb compensation | Day 1
  Limb compensation is a parameter calculated by the AuReha Web Platform that monitors any incorrect compensatory movements performed by the limbs during exercises. For example, it can detect shoulder elevation during elbow flexion, or elbow flexion during shoulder movements. This parameter is crucial for identifying and correcting dysfunctional movement patterns that could compromise the rehabilitation process.
  Unit of Measure: Percentage (%)
Characterization of AuReha in measuring the distance to a specified target | Day 1
  This parameter evaluates the final distance from the target to be reached. Unit of Measure: Percentage (%)
Characterization of AuReha in measuring the duration of the movement | Day 1
  This parameter calculates the duration of movement execution. Unit of Measure: seconds (s)
Characterization of AuReha in terms of usability for patients with the System Usability Scale (SUS) | Day 1
  Assessment of the usability of AuReha by enrolled patients during the evaluation and execution of proprioceptive exercises.
  Standardized questionnaires will be used (SUS). The questionnaire assesses usability and overall user experience. Responses are based on a 0-4 Likert difficulty scale (from "no difficulty" to "system unusable").
Characterization of AuReha in terms of usability for patients with the User Engagement Scale - Short Form (UES-SF) | Day 1
  Assessment of the usability of AuReha by enrolled patients during the evaluation and execution of proprioceptive exercises.
  Standardized questionnaires will be used (UES-SF). This questionnaire collects user feedback on the AuReha App and the sensorized shirt, focusing on the engagement. Responses are based on a 0-4 Likert difficulty scale (from "no difficulty" to "system unusable").
Characterization of AuReha in terms of usability for patients | Day 1
  Assessment of the usability of AuReha by enrolled patients during the evaluation and execution of proprioceptive exercises.
  Custom questionnaires have been developed for this purpose and are annexed to the clinical protocol. These questionnaires collect user feedback on the AuReha App and the sensorized shirt, focusing on usability, engagement, clarity of instructions, and garment fit. Responses are based on a 0-4 Likert difficulty scale (from "no difficulty" to "system unusable"), and include open-text fields for qualitative insights.
Characterization of AuReha in terms of usability for healthcare professionals | Day 1
  Standardized questionnaires will be used, specifically the Healthcare System Usability Scale (HSUS). In addition, custom questionnaires have been developed for this purpose and are annexed to the clinical protocol. These questionnaires collect user feedback on the AuReha App and the sensorized shirt, focusing on usability and clarity of instructions. Responses are based on a 0-4 Likert difficulty scale (from "no difficulty" to "system unusable") and include open-text fields for qualitative insights.
Correlation between AuReha shirt size (categorical: XS, S, M, L,) and the anthropometric measurements of healthy volunteers (in cm) | Day 1
  Evaluation of AuReha's fit on healthy volunteers, through the assessment of the correlation between the selected shirt size (categorical: XS, S, M, L) and continuous anthropometric variables, including body circumferences and segment lengths. Circumferences (in cm) will include: chest, waist, hips, upper arm, and forearm. Segment lengths (in cm) will include: shoulder to iliac spine and shoulder to wrist. All measurements will be taken using a standard anthropometric tape measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Poliambulatorio Shoulder Team, Forlì, FC, Italy

IPD SHARING:
Plan to Share IPD: Undecided